CLINICAL TRIAL: NCT02919358
Title: The Mozart Effect and the Assessment of Weight Gain and Development of Feeding Skills in the NICU.
Brief Title: Music and Feeding in NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DDD603441
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Feeding; NICU; Preterm Infants; Mozart; Weight Gain
MeSH Terms: conditions — Weight Gain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music (Experimental): Exposure to music, twice per day for the study period
  Interventions: Other: Music
- Control (Other): No intervention; standard care.
  Interventions: Other: No music.

INTERVENTIONS:
Other: Music
  Arms: Music
Other: No music. — This is the control group.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the effect of classical music exposure on improved time to regain birth weight and improved feeding readiness in healthy premature infants in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* • Neonates between the gestational ages of 28 weeks and 32 weeks and 6 days

  * Parents ≥18 years of age
  * English speaking parents
  * Breastmilk as intended primary form of nutrition

Exclusion Criteria:

* Congenital anomalies affecting hearing or feeding skills
* Patients requiring HFOV or HFJV

Ages: 28 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is time to regain birth weight | 2 weeks
  We will track weight gain and will monitor how long it takes for the babies to regain their birth weight.

SECONDARY OUTCOMES:
Assessment of Feeding Cues | 2 weeks
  At 33 weeks corrected gestational age; a speech therapist will assess feeding cues daily using an objective oral feeding assessment tool

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No